CLINICAL TRIAL: NCT01598480
Title: To Study the Healing Effect of Silver Impregnated Activated Carbon Fiber Wound Dressing on Superficial Dermal Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bio-medical Carbon Technology Co., Ltd. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201201004DSA
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Burns
Keywords: Burns; Wound Healing
MeSH Terms: conditions — Burns | interventions — Silver Sulfadiazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Flamazine is applied on the wound in the control group instead and then covered with sterile gauze.
  Interventions: Drug: Flamazine
- BCT Antimicrobial Dressing (Experimental): The wound in the experimental group is first cleansed with normal saline and then applied with BCT Antimicrobial Dressing and covered by sterile gauze, and dressings will be changed every 3 days.
  Interventions: Device: BCT Antimicrobial Dressing

INTERVENTIONS:
Drug: Flamazine — Silver sulfadiazine cream
  Arms: Control
Device: BCT Antimicrobial Dressing — Activated carbon fiber impregnated with silver particles
  Arms: BCT Antimicrobial Dressing

SUMMARY:
Background:

Bio-medical Carbon Technology (BCT) Antimicrobial Dressing, a novel advanced wound dressing invented by Bio-medical Carbon Technology Co., Ltd., Taiwan, consists principally of activated carbon fiber impregnated with silver particles. The highly porous nature and the large specific surface area of activated carbon fiber provide a tremendous adsorptive capacity for toxins, wound degradation products, and odors. Furthermore, far infrared ray emitted from activated carbon fiber accelerates blood circulation to stimulate tissue regeneration. Silver ions efficiently eliminate a broad spectrum of bacteria through penetrating the cell wall of bacteria and denaturing essential proteins. This clinical trial investigates wound healing effects of BCT Antimicrobial Dressing on superficial dermal burn patients.

Aim:

To investigate wound healing effects of BCT Antimicrobial Dressing on superficial dermal burn.

Methods:

This trial is expected to recruit 30 eligible subjects. After hospitalized patients are diagnosed as superficial dermal burn, the procedure of Informed Consent is conducted by the project investigator. As long as the patient agrees to join this clinical trial and signs the Informed Consent, two separate areas of 25 cm2 in the same anatomic site are chosen and distributed to the control and research groups respectively by coin flipping. The wound in the research group is first cleansed with normal saline and then applied with BCT Antimicrobial Dressing and covered by sterile gauze, and dressings will be changed every 3 days (counting from the day applied BCT dressings: Day0, 3, 6, 9, 12, 15……etc.) until the wound is healed. Flamazine is applied on the wound in the control group instead and then covered with sterile gauze, and the frequency of dressing change is daily until the wound is recovered. The healed and non-healed area of wound is recorded and photographed every 3 days, and the wound color and infection are also evaluated. On Day 12 and Day 21, compare the ratio of healing and non-healed areas in the control and research groups, and the ending point is set on the 21st day.

Statistics Analysis:

Paired Student's t-test will be performed to analyze the clinical data by comparing the difference of the healing percentage, the healing rate, the infection rate, and the frequency of dressing change. It is statistically significant when P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* The total burn area is between 5% to 30%
* Male/Female of any race aged between 20 - 80 years old
* Non taking any medicine containing steroid
* No allergy to activated carbon fiber and silver
* No history of cardiovascular diseases, diabetes mellitus, immune system-related diseases, hepatic disease, hematic diseases, renal diseases, and cancer

Exclusion Criteria:

* The total burn area is less than 5% or larger than 30%
* Male/Female of any race aged younger than 20 years old or older than 80 years old
* Taking any medicine containing steroid
* Allergy to activated carbon fiber and silver
* With history of cardiovascular diseases, diabetes mellitus, immune system-related diseases, hepatic disease, hematic diseases, renal diseases, and cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The healing rate | 21 days
  Photograph of wounds are taken on the specific day (Day0, 3, 6, 9……etc.) and pictures are imported to image-analyzing software for the calculation of wound area. And the number of wound area is then transformed to the healing percentage and the healing rate. Healing Rate= healed area/the number of healing days (cm2/day)

SECONDARY OUTCOMES:
The healing percentage | 21 days
  Photograph of wounds are taken on the specific day (Day0, 3, 6, 9……etc.) and pictures are imported to image-analyzing software for the calculation of wound area. And the number of wound area is then transformed to the healing percentage. Healing Percentagen =[(the initial wound area-wound area measured on Dayn)/the initial wound area]x100%. N means the number of days counting from the first day initiating this clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Eng Kean Yeong, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Burn Center, Department of Surgery, National Taiwan University Hospital, Taipei, Taiwan